CLINICAL TRIAL: NCT06551584
Title: Phase I Trial for Patients With Advanced Hematologic Malignancies Undergoing Allogeneic Hematopoietic Cell Transplantation From an HLA-Mismatched Donor (7/8) With Orca-T
Brief Title: Phase I Trial for Patients w/ Advanced Hematologic Malignancies Undergoing Allogeneic HCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-73393; NCI-2025-01029 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Mixed Phenotype Acute Leukemia; Myelodysplastic Syndromes
Keywords: Orca-T; Hematopoietic Cell Transplantation; Advanced Hematologic Malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ORCA-T + (tacrolimus and ruxolitinib) (Experimental): Dual-agent tacrolimus starting on the day after Tcon infusion (Day +3 or Day +4) and ruxolitinib starting on the day after tacrolimus (Day +4 or Day +5).
  Interventions: Drug: ORCA-T

INTERVENTIONS:
Drug: ORCA-T — On Day 0, participants will receive an infusion of Orca-T HSPCs and Orca-T Tregs. On Day +2 or +3 (between approximately 48 to 72 hours of Day 0), patients will receive an infusion of the Orca-T Tcons. There is no dose escalation or de-escalation planned for the Orca-T investigational product.

SUMMARY:
The study goal is to characterize the safety of the combination of Orca-T with dual agent GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible diseases:

   * Acute myeloid, lymphoid or mixed phenotype leukemia in complete remission (CR) or CR with incomplete hematologic recovery (CRi) as defined in Section 6.1.3; with or without the presence of known minimal residual disease, or
   * Myelodysplasic syndrome (MDS) myelodysplastic syndromes eligible for alloHSCT and/or treatment-related MDS <10% blasts
2. Age ≥ 18 and ≤ 70 years at the time of enrollment.
3. Eligible for myeloablative alloHCT including one of two the myeloablative conditioning regimens (fractionated total body irradiation plus cyclophosphamide or busulfan, fludarabine, and thiotepa)
4. Has a related or unrelated donor available who is 7/8 match (single allele mismatched) at HLA-A, -B, -C, and -DRB1, all typed using DNA-based high-resolution methods.
5. Estimated glomerular filtration rate (eGFR) ≥ 50 mL/minute or creatinine < 2 mg/dL.
6. Cardiac ejection fraction at rest ≥ 45% or shortening fraction of ≥ 27% by echocardiogram or radionuclide scan (MUGA).
7. Diffusing capacity of the lung for carbon monoxide (DLCO) (adjusted for hemoglobin) ≥ 50%.
8. Total bilirubin < 2 times upper limit of normal (ULN) (patients with Gilbert's syndrome may be included once hemolysis has been excluded).
9. Ability to understand and the willingness to provide written informed consent.
10. Negative serum or urine beta-HCG test in females of childbearing potential (FCBP) within 3 weeks of enrollment.

    A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
11. Able to give informed consent. Legal authorized representative (LAR) is permitted if subject is cognitively able to provide verbal assent.
12. Karnofsky Performance Score ≥70%

Exclusion Criteria:

1. Prior allogeneic HCT.
2. Currently receiving corticosteroids or other immunosuppressive therapy. Topical corticosteroids or oral systemic corticosteroid doses less than or equal to 10 mg/day are allowed.
3. Planned donor lymphocyte infusion (DLI).
4. Planned pharmaceutical in vivo or ex vivo T cell depletion, e.g., post-transplant cyclophosphamide (Cy), peri-transplant anti-thymocyte globulin (ATG), or alemtuzumab. For patients that have previously been exposed to a T cell-depleting agent, a 5 half-life washout of the agent must occur prior to planned Day 0 (day of infusion of Orca-T HSPC and Tregs ).
5. Recipient positive anti-donor HLA antibodies against a mismatched allele in the selected donor determined by either:

   1. Positive crossmatch test of any titer (by complement-dependent cytotoxicity or flow cytometric testing), or
   2. Presence of anti-donor HLA antibody to any of the following HLA loci: HLA-A, -B, -C, -DRB1, -DQB1, -DQA1, -DPB1, or -DPA1, with mean fluorescence intensity (MFI) >1000 by solid phase immunoassay.
6. Uncontrolled bacterial, viral, or fungal infections (currently taking antimicrobial therapy and with progression or no clinical improvement) at time of enrollment including known, active tuberculosis infection.
7. Seropositive for HIV-1 or -2, HTLV-1 or -2, Hepatitis B sAg, and/or Hepatitis C antibody.

   *History of hepatitis B or hepatitis C is permitted if viral load is undetectable per quantitative PCR and/or NAT. In this case, monitoring for hepatitis B or hepatitis C by PCR at 3, 6, and 12 months is recommended.
8. Known allergy or hypersensitivity to, or intolerance of, any investigational agent or ingredient therein, or planned GVHD prophylactic medications.
9. Documented allergy or hypersensitivity to iron dextran or bovine, murine, algal or Streptomyces avidinii proteins.
10. Any uncontrolled autoimmune disease requiring active immunosuppressive treatment.
11. Concurrent malignancy diagnosed within 12 months of enrollment, except non-melanoma skin cancers that have been curatively resected.
12. Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use effective forms of birth control or abstinence for one year after transplantation.

    (FCBP definition: A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
13. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment. History of stroke or pulmonary embolism within 6 months of enrollment.
14. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the recipient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Without Severe Transplant-Related Adverse Events at Day +100 | 18 months
  The proportion of patients who, at Day +100 have not experienced any severe transplant-related adverse events including non-relapse mortality (NRM), primary graft failure, acute GVHD (grade 2-4), acute GVHD grade 3-4, or opportunistic infections (grade 4-5).

CONTACTS AND LOCATIONS:
Overall Officials: Lori Muffly, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States